CLINICAL TRIAL: NCT01634880
Title: Phase II Trial of Postoperative Radiotherapy and Panitumumab in High-Risk Salivary Gland Malignancies
Brief Title: Postoperative Radiotherapy and Panitumumab in High-Risk Salivary Gland Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual.
Sponsor: Athanassios Argiris (Other)
Collaborators: University of Pittsburgh (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Athanassios Argiris, Principal Investigator, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRC 11-37; HSC20120130H (Other: UTHSCSA IRB)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Salivary Gland Malignancy
Keywords: Salivary Gland Malignancies; Panitumumab; Postoperative; Radiotherapy
MeSH Terms: interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Postoperative Radiotherapy and Panitumumab (Experimental)
  Interventions: Drug: Postoperative Radiotherapy and Panitumumab

INTERVENTIONS:
Drug: Postoperative Radiotherapy and Panitumumab — The starting panitumumab dose is 2.5 mglkg given once a week. The total dose may be rounded up or down by no greater than 10 mg. The panitumumab dose will be calculated based on the subject's actual weekly body weight.
  Standard radiation 64-70Gy with 2.0 Gy daily fractions in 6-7 weeks. Panitumumab 2.5 mg/Kg IV, weekly during radiation (total of 6-7 doses).

SUMMARY:
Standard therapy for high-risk or locally advanced salivary gland malignancies is surgery followed by postoperative radiation therapy. Studies have shown the superiority of combined modality therapy compared to surgery alone. Despite the addition of postoperative radiation therapy, the five-year survival for locally advanced salivary gland malignancies is poor (less than 60%). In salivary gland malignancies, the epidermal growth factor receptor (EGFR) is expressed in 25-85%; in certain histological types, like salivary duct carcinomas, the expression is higher. EGFR is a promising target of anticancer therapy. In squamous cell carcinoma of the head and neck, a phase III trial utilizing cetuximab added to radiation therapy improved both locoregional control and overall survival compared to radiation alone. Panitumumab is a novel, human, IgG2 EGFR monoclonal antibody that may be better tolerated and more efficacious than cetuximab. Here, the investigators hypothesize that the addition of panitumumab to standard radiotherapy in locally advanced salivary gland malignancies will improve recurrence-free survival (RFS).

DETAILED DESCRIPTION:
Specific Aims To determine the recurrence-free survival (primary endpoint), overall survival, local and distant recurrence-free survival, and treatment-related toxicities. Also, the investigators plan to study EGFR-related and immune biomarkers in baseline tumor tissue as well as blood samples obtained prior and after therapy.

Subject Population We will enroll patients with completely resected, locally advanced salivary gland cancers.

Treatment Plan Standard radiation 64-70Gy with 2.0 Gy daily fractions in 6-7 weeks. Panitumumab 2.5 mg/Kg IV, weekly during radiation (total of 6-7 doses).

Statistical Design and Sample Size Phase II, one-stage, study with the 3-year recurrence-free survival (RFS) as the primary endpoint. The sample size is 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically determined salivary gland cancer of the major or minor salivary glands of the head and neck (any histology) status post potentially curative surgical resection with no macroscopic residual disease. Patients should have AJCC 6th edition stage III with 1) extracapsular extension, 2) perineural invasion, 3) positive surgical margins or 4) high grade histology or stage IVA or IVB.
* No distant metastasis.
* No prior chemotherapy, biological-targeted therapy (including any prior therapy which specifically and directly targets the EGFR pathway), or radiotherapy for head and neck cancer.
* No more than 10 weeks (minimum of 3 weeks) should elapse between surgery and treatment on study.
* ECOG performance status of 0-2.
* Patients must have normal organ and marrow function.
* No prior invasive malignancy unless the disease-free survival is 3 years or more.
* Age 18+ years.
* Pregnant or breast-feeding women are excluded (see exclusion criteria).
* Informed consent must be obtained from all patients prior to beginning research related treatment.
* Patients should have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months) uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction. All patients will have a baseline EKG. If abnormalities consistent with active coronary artery disease are detected, the patient will be referred to a cardiologist for appropriate evaluation and management prior to treatment on study.
* Patients may not be receiving any other investigational agents.
* No history of prior malignancy, with the exception of basal carcinoma of the skin or in situ cervical cancer, or malignancy that has been treated with a curative intent with a 3-year disease-free survival.
* Pregnant women are excluded from this study because chemotherapy and radiation therapy have the potential for teratogenic or abortifacient effects.
* All WOCBP must have a negative serum pregnancy test at baseline, or within 7 days prior to receiving investigational product. All WOCBP should be instructed to contact the Investigator if they suspect they might be pregnant.
* Prior severe infusion reaction to a human monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival | 5-7 years
  To evaluate the recurrence-free survival of locoregionally-advanced (stages III/IV) salivary gland cancer patients undergoing postoperative chemoradiotherapy with panitumumab compared to historical control data. Survival measured by RECIST criteria and analyzed using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Overall survival | 5-7 years
  Overall survival will be measure via RECIST criteria and analyzed using the Kaplan-Meier method.
Efficacy | 5 years
  Correlate efficacy parameters with EGFR and downstream pathway activation,FcyR polymorphisms, and serum cytokine profiles. More specifically, the aim is to demonstrate the usefulness of biomarkers (downstream signaling molecules, FcyR polymorphisms, or tumor and serum cytokine(s) in predicting recurrence-free survival in patients with salivary gland cancer treated with the above treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas, United States